CLINICAL TRIAL: NCT04348487
Title: Modified Cephalica Venous Access Port Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Putu Anda Tusta Adiputra, Consultant, Division of Surgical Oncology, Department of Surgery, Udayana University, Udayana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UdayanaU
Record Dates: First submitted 2018-11-18; First posted 2020-04-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Chemotherapy Effect; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Introducing new approach of chemoport insertion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard procedure (Other): For the conventional TIVAPS with cephalic vein approach, incision was made either in the midline of infraclivular or supraclavicular. Cathether was introduced to the central and then connected to the laterally implanted port in the deltopectoral region. The experience in the local center experienced several pitfalls with this method such as pneumothorax, pinch-off syndrome, compression of the catheter by the clavicle, kinking of the catheter, and loss of patencty.
  Interventions: Other: Modified cephalica venous access

INTERVENTIONS:
Other: Modified cephalica venous access — This modified technique prioritized the safety in TIVAPS by using several modified landmarks and techniques. The catheter was inserted through cephalic vein in deltopectoral groove regio and implanted the port in the anteromedial of thorax. Generally, the percutaneous and Seldinger technique was used to ensure safety and minimal tissue disruption. To connect the trimmed catheter to port pocket, the author anchored a special trocar from anteromedial of thorax to the deltopectoral groove for guidance.

SUMMARY:
As long term totally implantable central venous access (TIVAPS) was increasingly needed in cancer patient, some modified techniques were introduced to improved the outcome and safety of the port implantation. In this modified technique, the prioritization were the safety and stability of catheter and port placement. Catheter was inserted to the cephalic vein in the deltopectoral groove, in which connected to the port pocket implanted in the anteromedial thorax. Connection was done by percutaenous and Seldinger technique by introducing a special trocar to ensure safety. Long term outcome was satisfactorily good by this technique without and major and minor events.

DETAILED DESCRIPTION:
Large studies have proved that TIVAPS was effective for long term venous access with minimal risk of complication. For TIVAPS, clinicians have approach the vena cava through the subclavian, internal jugular vein, or cephalic vein regularly with various technique. The most minimal complication risk was obtained in the access through cephalic vein.In the conventional method of cephalic central venous access approach, the incision was done at clavicular regio, with the high risk of catheter being kinking. To improve the feasibility of the techique, here, the author introduced the modified technique for cephalic vein approach.

Step 1 Preparation The patient was positioned supine with the head tilted to the left. In our procedure, the head was tilted to the left in order to expose the deltopetoral groove. The procedure was done in aseptic condition with iodine tincture and sterile draping. It was carried out under local anesthesia in an operating room. A two-gram of cephazolin was inserted intravenously following the guideline standard in the local hospital.

Step 2 Landmarks There were two landmark incision in this procedure, in which the first one is in deltopectoral groove for catheter insertion and the second is in anteromedial of thorax. The deltopectoral groove is located between the insertio of pectoralis major and deltoid muscle. The cephalic vein passes through the clavipectoral (deltopectoral) triangle to join the axillary vein. Lidocaine without adrenaline was used as a local anesthetic in both incision. The procedure was done without any radiology guidance.

Step 3 Vein identification The first incision was made for the insertion of venous catheter. As long as 2 to 3 cm incision was made in the deltopectoral groove. An incision of 3 mm in length was made on the surface of the vein. The incision was then deepened to the fascia overlying the deltoid and pectoralis muscle. Subcutaneous tissue was positioned by blunt dissection to uncover the cephalic vein. The cephalic vein was identified in the adipose tissue along the deltopectoral groove. Surgical cauterization was used to control bleeding. The proximal and distal end of the vein was secured by tying and a hemostat was applied for traction. A transverse venotomy was made at the center of these 2 sutures.

Step 4 Venous catheter insertion A peel-away sheath was inserted to facilitate the catheter insertion into the venous system. The catheter was inserted into the cephalic vein for approximately 25 centimeters.

Step 5 Port pocket incision The 3-4 cm for second incision was carried out for port pocket, with the position on anteromedial of thorax for chemoport implantation. Trocar was tunneled subcutaenously and advanced to the first incision. Catheter was trimmed and ready to be connected to the reservoir.

Step 6 Port implantation The port was inserted to the port pocket and anchored to two sites of underlying muscle in chest was using permanent monofilament suture. The implanted port was flushed with 10 ml of normal saline and 5 ml of 50 IU/ml heparin.

Step 7 Ensuring position For ensuring the catheter position, plain chest radiograph (posteroanterior view) was done.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are planning to receive chemotherapy and need chemoports placement.

Exclusion Criteria:

* Unconsented subjects

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
patency of chemoport | 10 minutes after the insertion of chemoport
  While flushing 10 ml of saline to chemoport, measure the velocity flow of saline injection. If the saline was complete in less than 1 minute, it was considered normal. difficulty in flushing the chemoport and pain during flushing should be considered as a failure.
location of chemoport | 1 hour after the insertion of chemoport.
  appropriate location of chemoport can be found by thorax X Ray, confirmed by radiographers evaluation.

SECONDARY OUTCOMES:
complication of chemoport | 1 month after the insertion of chemoport
  observation any sign of infection

CONTACTS AND LOCATIONS:
Overall Officials: Putu Anda Tusta Adiputra, MD, Principal Investigator — Division of Surgical Oncology, Department of Surgery, Udayana University
Locations (1):
- Putu Anda Tusta Adiputra, Denpasar, Bali, Indonesia